CLINICAL TRIAL: NCT06749951
Title: Cognitive Behavioural Therapy for Insomnia in Patients With Coronary Heart Disease: A Randomized Controlled Trial With Six Months Follow-up
Brief Title: Cognitive Behavioural Therapy for Insomnia in Patients With Coronary Heart Disease
Acronym: TreatSleepCHD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vestre Viken Hospital Trust (Other)
Collaborators: Oslo University Hospital (Other); University of Oslo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 678911
Record Dates: First submitted 2024-12-11; First posted 2024-12-27 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Insomnia Chronic; Coronary Heart Disease
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Coronary Disease | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Behavioural Therapy for insomnia (CBT-I) (Experimental)
  Interventions: Other: Cognitive Behavioural Therapy for insomnia (CBT-I)
- Sleep Hygiene Advice (Active Comparator)
  Interventions: Other: Sleep Hygiene Advice

INTERVENTIONS:
Other: Cognitive Behavioural Therapy for insomnia (CBT-I) — Five 60-90 minutes weekly sessions delivered by an appropriately trained cardiac nurse at a cardiology department. The CBT-I intervention will follow a manualized treatment protocol developed by Espie and colleagues (Espie et al. 2001, 2007, 2008) and evaluated in a number of published RCTs using CBT-I. The key components of this intervention include sleep hygiene advice, stimulus control, sleep restriction, relaxation training, and cognitive restructuring.
  Arms: Cognitive Behavioural Therapy for insomnia (CBT-I)
Other: Sleep Hygiene Advice — "Sleep well" is a 16-page written brochure developed by the Directorate of Health in Norway for dissemination to patients with sleep problems including insomnia. It covers general sleep hygiene advice (setting a regular bed-time, avoiding stimulants, alcohol and exercise in the evening, sleeping in a quiet bedroom, advice of practicing relaxation technique and postpone worries).
  Arms: Sleep Hygiene Advice

SUMMARY:
Insomnia is prevalent (45%) in CHD patients and associated with significantly increased risk for recurrent cardiovascular events. Insomnia has recently been identified as the third most important risk factor for prognosis. However, very few insomnia patients are identified and receive treatment of insomnia today. CBT-I is the first-line treatment for insomnia, but studies on the effects in CHD patients are lacking. This project aims to document the effectiveness of Cognitive Behavioural therapy for insomnia (CBT-I) in an outpatient population with coronary heart disease (CHD). Furthermore, the biological and psychological mechanisms that may mediate the effects of the intervention will be identified. Finally, a health-economic simulation and a qualitative study of the participants experiences with CBT-I will be performed. This prospective, randomized, intervention study will continue until data have been collected for the primary outcome on 66 CHD outpatients with a diagnosis of insomnia assessed by Bergen Insomnia Scale (BIS). Participants will be randomised to a short, nurse-administered, CBT-I delivered in a group format or to sleep hygiene advice. The primary outcome will be remission from BIS-insomnia post-treatment and at 6-months follow-up. Secondary outcomes will be changes in insomnia severity, objective and subjective sleep parameters, daytime symptoms of insomnia, and quality of life. Exploratory outcomes include inflammation, cortisol, HbA1C, and cognitions/metacognitions. The project may document the effectiveness of CBT-I for a large patient-group with potentially favorable long-term effects on important clinical outcomes.

ELIGIBILITY:
Inclusion criteria (all the following):

* Aged 18-75 years and signed informed consent and expected cooperation according to ICH/GCP and national/local regulations
* Hospitalised with acute myocardial infarction and/or angiography-verified coronary atherosclerosis, or a coronary revascularisation procedure at Drammen Hospital 2021-2024
* A positive score for insomnia measured with Bergen Insomnia Score
* At least 10 of 14 daily diaries completed of the sleep diary during pre-randomization assessment

Exclusion criteria (any of the following):

* Any condition or situation, that in the investigator's opinion could put the subject at significant risk, confound the study results, interfere significantly with the subject participation in the study, or rendering informed consent unfeasible not limited to:
* Moderate or severe cognitive impairment (i.e. recorded in hospital records or a Montreal Cognitive Assessment brief version score < 11), seizure disorders, active suicidal intent or plans, substance or alcohol dependence, psychotic disease, major depressive disorders or bipolar disorders, receiving concurrent psychological treatments, and ongoing night shift work.
* Neurological or musculoskeletal disorders that restrict movement of the dominant arm because of the possible confounding effects on wrist actigraphy recordings.
* A diagnosis of heart failure recorded in the hospital medical records and/or an NT-proBNP >125 pg/mL
* Short life expectancy (<12 months) due to end-organ (i.e COPD 4, CKD 4/5) or malignant diseases
* Not being able to understand Norwegian.
* No other significant sleep disorder, as assessed via the Structured Clinical Interview for Sleep disorders (Kallestad et al., 2022)
* A clinical diagnosis of Obstructive Sleep Apnea (OSA) (not treated with CPAP) recorded in the hospital medical records, under evaluation for OSA, and/or a score ≥5 on the STOP-Bang OSA screening questionnaire

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2024-12-30 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Remission clinical diagnosis of insomnia | From baseline to weeks 6-8 and 26
  Between- and within- group differences in the proportion witn remission of insomnia diagnosis assessed by the Bergen Insomnia Scale
Changes in insomnia severity | From baseline to weeks 6-8 and 26
  Between- and within- group differences in insomnia severity assessed by the Insomnia Severity Index

SECONDARY OUTCOMES:
Changes in insomnia assessed by the Pittsburgh Sleep Quality Index | From baseline to weeks 6-8 and 26
  Between- and within- group differences in insomnia assessed by the Pittsburgh Sleep Quality Index with higher scores indicating worse outcomes
Changes in subjective sleep efficiency | From baseline to weeks 6-8 and 26
  Between- and within- group differences in sleep efficiency assessed by a self-report sleep diary with higher scores indicating better outcomes
Changes in objective sleep efficiency | From baseline to weeks 6-8 and 26
  Between- and within- group differences in sleep efficiency assessed by an assessed by an actigraph with higher scores indicating better outcomes
Changes in subjective total sleep time | From baseline to weeks 6-8 and 26
  Between- and within- group differences in total sleep time assessed by a self-report sleep diary with higher scores indicating better outcomes
Changes in objective total sleep time | From baseline to weeks 6-8 and 26
  Between- and within- group differences in total sleep time assessed by an assessed by an actigraph with higher scores indicating better outcomes
Changes in subjective sleep onset latency | From baseline to weeks 6-8 and 26
  Between- and within- group differences in sleep onset latency assessed by a self-report sleep diary with higher scores indicating worse outcomes
Changes in objective sleep onset latency | From baseline to weeks 6-8 and 26
  Between- and within- group differences in sleep onset latency assessed by an assessed by an actigraph with higher scores indicating worse outcomes
Changes in subjective wake after sleep onset | From baseline to weeks 6-8 and 26
  Between- and within- group differences in wake after sleep onset assessed by a self-report sleep diary with higher scores indicating worse outcomes
Changes in objective wake after sleep onset | From baseline to weeks 6-8 and 26
  Between- and within- group differences in wake after sleep onset assessed by an assessed by an actigraph with higher scores indicating worse outcomes
Changes in symptoms of depression and anxiety | From baseline to weeks 6-8 and 26
  Between- and within- group differences in symptoms of depression and anxiety assessed by the Hospital and Anxiety Depression Scale with higher scores indicating worse outcomes
Changes in daytime sleepiness | From baseline to weeks 6-8 and 26
  Between- and within- group differences in daytime sleepiness assessed by the Epworth Sleepiness Scale with higher scores indicating worse outcomes
Changes in fatigue | From baseline to weeks 6-8 and 26
  Between- and within- group differences in fatigue assessed by the Chalder Fatigue Scale with higher scores indicating worse outcomes
Changes in general quality of life | From baseline to weeks 6-8 and 26
  Between- and within- group differences in quality of life assessed by the 5-level EQ-5D version with higher scores indicating better outcomes
Changes in sleep-related quality of life | From baseline to weeks 6-8 and 26
  Between- and within- group differences in sleep-related quality of life assessed by the Glasgow Sleep Impact Scale with higher scores indicating better outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- Vestre Viken Trust Drammen hospital, Drammen, Buskerud, Norway